CLINICAL TRIAL: NCT04848584
Title: Pfizer-BioNTech COVID-19 BNT162b2 Vaccine Effectiveness Study - Kaiser Permanente Southern California
Brief Title: Pfizer-BioNTech COVID-19 Vaccine Effectiveness Study - Kaiser Permanente Southern California
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591014; NCT04848584 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-03-30; First posted 2021-04-19 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Fully vaccinated: Prior receipt of 2 doses of BNT162b2 received with ≥7 days between receipt of the 2nd dose and the index date. This group will serve as the 'exposed' group evaluated in the primary objective.
  Interventions: Biological: Primary Exposure Status of Pfizer-BioNTech COVID-19 Vaccine; Biological: BNT162b2 BA.4/5 bivalent
- Partially vaccinated: Prior receipt of 1 dose (only) of BNT162b2 received with ≥14 days between receipt of the 1st dose and the index date.
  Interventions: Biological: Primary Exposure Status of Pfizer-BioNTech COVID-19 Vaccine; Biological: BNT162b2 BA.4/5 bivalent
- Ever vaccinated: Prior receipt ≥1 dose of BNT162b2 received with ≥14 days between index date and receipt of the 1st dose
  Interventions: Biological: Primary Exposure Status of Pfizer-BioNTech COVID-19 Vaccine
- Never vaccinated: never received BNT162b2. This group will serve as the reference exposure group (i.e., 'unexposed' group) in all VE analyses
  Interventions: Biological: Primary Exposure Status of Pfizer-BioNTech COVID-19 Vaccine; Biological: BNT162b2 BA.4/5 bivalent
- Bivalent vaccinated: Receipt of the BNT162b2 BA.4/5 bivalent vaccine ≥8 weeks (≥56 days) since the most recent dose of wild-type COVID-19 mRNA vaccine (BNT162b2 or mRNA-1273) received
  Interventions: Biological: BNT162b2 BA.4/5 bivalent
- XBB.1.5 vaccinated: Receipt of XBB.1.5-adapted monovalent vaccine with greater than or equal 14 days between receipt of vaccine and the event date.
  Interventions: Biological: XBB.1.5-adapted vaccinated
- Unexposed to XBB.1.5: Unvaccinated with XBB.1.5-adapted monovalent vaccine or any other manufacturer's XBB-adapted formulation.
  Interventions: Biological: XBB.1.5-adapted vaccinated

INTERVENTIONS:
Biological: Primary Exposure Status of Pfizer-BioNTech COVID-19 Vaccine — prior administration of Pfizer-BioNTech COVID-19 vaccine; vaccine is not administered in this study
  Other Names: COVID VACCINE
  Groups: Ever vaccinated; Fully vaccinated; Never vaccinated; Partially vaccinated
Biological: BNT162b2 BA.4/5 bivalent — Vaccination with a bivalent booster was defined as receipt of the BNT162b2 BA 4/5 bivalent vaccine ≥8 weeks (≥56 days) since the most recent dose of wild-type COVID-19 mRNA vaccine (BNT162b2 or mRNA-1273) received.
  Groups: Bivalent vaccinated; Fully vaccinated; Never vaccinated; Partially vaccinated
Biological: XBB.1.5-adapted vaccinated — Vaccinated with XBB.1.5-adapted vaccine
  Groups: Unexposed to XBB.1.5; XBB.1.5 vaccinated

SUMMARY:
The primary objective of this study is to determine the vaccine effectiveness of 2 doses of Pfizer-BioNTech BNT162b2 vaccine against COVID-19-associated hospitalization. There will be a large retrospective database study using two parallel study designs: a test-negative case-control design and a retrospective cohort design. VE estimates by various strata and strain type will be conducted.

DETAILED DESCRIPTION:
The primary objective of the study is to estimate vaccine effectiveness (VE) of 2 doses of Pfizer's BNT162b2 vaccine against acute respiratory illness (ARI) requiring hospitalization due to SARS-CoV-2 infection among KPSC members eligible for vaccination. VE will be evaluated using a test-negative design (TND), including all KPSC patients eligible for vaccination who are admitted to the hospital with (ARI) after 14 December 2020 (date of first vaccinations at KPSC), and who receive a PCR test for SARS-CoV-2. Secondary and exploratory objectives may examine VE for 1 dose vaccination, at least 1 dose, >2 doses, monovalent, bivalent or mixed dosing schedules as well as against ED admission, specific variants, mixed dosing schedules, durability, age cut-offs to align with regulatory authorizations/approvals and other populations of interest. Additionally, we will estimate VE using a full cohort design, including all KPSC members eligible for vaccination.

To assess VE, we propose a large retrospective database study using two parallel study de-signs: a test-negative case-control design and a retrospective cohort design. The TND will assess VE against COVID-19 hospitalization (primary endpoint) and ED admission. The retrospective cohort analysis may assess VE against COVID-19 hospitalization (primary), ICU admission, death, ED admission, and outpatient disease (with no subsequent hospitalization within 14 days). The BNT162b2 BA.4/BA.5 bivalent vaccine effectiveness will only be assessed via a test negative design due to the limitations regarding testing bias. As the pandemic evolved PCR-confirmed testing and reporting became less routine and differences in health care seeking behaviors were seen based on vaccination status.

VE for the XBB1.5-adapted monovalent vaccine will be defined as receipt of Pfizer -BioNTech XBB1.5-adapted monovalent vaccine with greater than or equal to 14 days between receipt of vaccine and the event date.

We will further conduct additional analyses of VE estimates by various patient characteristics and strain types.

ELIGIBILITY:
Inclusion Criteria for Test Negative Design

* KPSC patients eligible to receive BNT162b2 who are admitted to the hospital (primary objective and some secondary objectives) with acute respiratory infection (ARI; International Classification of Diseases (ICD) codes) after 14 December 2020 (date of first vaccinations at KPSC), and who receive a PCR test for SARS-CoV-2.
* For secondary objectives estimating VE against ED admission, the TND will include KPSC patients eligible to receive BNT162b2 who present to the ED with ARI after 14 December 2020, and who receive a PCR test for SARS-CoV-2.
* We will include membership requirement of 1 year prior to index date, which is defined as the date of hospitalization or ED admission (allowing 31-day administrative gap), to facilitate accurate capture of comorbid conditions.

Inclusion Criteria for Cohort Design-

* All KPSC members as of 14 December 2020 (date of first Pfizer vaccination at KPSC) eligible to receive BNT162b2.
* For the cohort study, patients must have at least 1 year of membership (allowing 31-day administrative gap) prior to 14 December 2020 (index date, date vaccinations first began at KPSC) to facilitate accurate capture of comorbid conditions.

Exclusion Criteria Test Negative Design Patients who receive only another newly licensed or investigational SARS-CoV-2 vaccine or COVID-19 prophylactic agent other than Pfizer's COVID-19 vaccine prior to hospitalization (or ED, for secondary objective) will be excluded from the study population When estimating VE for BNT162b2 vaccination, patients receiving another newly licensed or investigational SARS-CoV-2 vaccine or COVID-19 prophylactic agent other than Pfizer's COVID-19 vaccine prior to hospitalization or ED will be excluded from the analysis. Patients will also be excluded if the index date is within certain time windows from vaccination date, outlined further in the exposure section below.

Exclusion Criteria for Cohort Design There will be no exclusion criteria for the cohort design, however patients will be censored for receiving any other newly licensed or investigational SARS-CoV-2 vaccine or COVID-19 prophylactic agent other than Pfizer's COVID-19 vaccine

XBB.1.5-adapted monovalent vaccine eligibility analyses:

Inclusion Criteria:

* KPSC membership for a minimum of 1 year prior to index date, allowing a 30-day gap in membership to allow for delays in renewal. Participants <1 year did not have a membership requirement.≥6 months of age as of index date
* Admitted to the hospital or had an encounter in the ED, UC, or OP setting with a diagnosis of acute respiratory infection (ARI; defined based on International Classification of Diseases (ICD) codes listed in Appendix Table 1) after 25 September 2023
* Received a SARS-CoV-2 PCR or rapid antigen test

Exclusion criteria:

* Individuals who received a non-Pfizer-BioNTech XBB.1.5-adapted monovalent vaccine
* Individuals with an index event <14 days after vaccination with Pfizer-BioNTech XBB.1.5-adapted monovalent vaccine
* Individuals receiving a mRNA bivalent BA4.5 booster ≤ 8 weeks (≤ 56 days) since receiving last wild type dose
* Individuals with <28 days between a second and subsequent wild type dose
* Individuals receiving a XBB.1.5-adapted monovalent vaccine ≤ 8 weeks (≤ 56 days) since receiving a mRNA bivalent BA4.5 booster
* Individuals receiving oral COVID-19 antiviral OP treatments within 30 days of index event (will be excluded for primary analysis, but included in sensitivity analyses)

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All members of KPSC who are eligible based on vaccination status and age.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Test Negative Design Outcome: VE calculated as 1 minus the odds ratio (OR) comparing the odds of being vaccinated with 2 doses with BNT162b2 for hospitalized cases and controls, multiplied by 100%. | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against hospitalization for Acute Respiratory Infection due to SARS-CoV-2 infection
Cohort Design Outcome: VE calculated as 1 minus the hazard ratio (HR) comparing the incidence of 2 doses with BNT162b2 for hospitalization due to SARS-CoV-2 infection and not, multiplied by 100%. | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against hospitalization due to SARS-CoV-2 infection
VE of XBB.1.5-adapted monovalent vaccine against hospitalization | up to three years
  chart reviews focused on the identification of hospitalizations that are clearly not for COVID-19.
VE of XBB.1.5-adapted monovalent vaccine against critical illness | up to three years
  Chart confirmed COVID-19 related to critical illness (death, mechanical ventilation, ICU)
VE of XBB.1.5-adapted monovalent against outpatient visits | up to three years
  Number of patients with identified acute respiratory illness (ARI) diagnosis
VE of XBB.1.5-adapted monovalent vaccine against UC/ED visits. | up to three years
  Number of patients with identified acute respiratory illness (ARI) diagnosis

SECONDARY OUTCOMES:
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of being vaccinated with 2 doses BNT162b2 for ED cases and controls, multiplied by 100% | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against ED admission (without subsequent hospitalization) for ARI due to SARS-CoV-2 infection
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of being partially vaccinated with BNT162b2 (only 1 dose) for hospitalized cases and controls, multiplied by 100%. | up to three years
  To describe the effectiveness of only 1 dose of BNT162b2 (i.e., partially vaccinated) against hospitalization for ARI due to SARS-CoV-2 infection.
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of being partially vaccinated with BNT162b2 (only 1 dose) for ED cases and controls, multiplied by 100%. | up to three years
  To describe the effectiveness of only 1 dose of BNT162b2 (i.e., partially vaccinated) against ED admission (without subsequent hospitalization) for ARI due to SARS-CoV-2 infection
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of ever being vaccinated (≥1 dose) with BNT162b2 for hospitalized cases and controls, multiplied by 100%. | up to three years
  To describe the effectiveness of ≥1 dose of BNT162b2 (i.e., ever vaccinated) against hospitalization for ARI due to SARS-CoV-2 infection
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of ever being vaccinated (≥1 dose) with BNT162b2 for ED cases and controls, multiplied by 100%. | up to three years
  To describe the effectiveness of ≥1 dose of BNT162b2 (i.e., ever vaccinated) against ED admission (without subsequent hospitalization) for ARI due to SARS-CoV-2 infection
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of >2 doses with BNT162b2 for hospitalized cases and controls, multiplied by 100%. | up to three years
  To describe the effectiveness of >2 doses of BNT162b2 against hospitalization for ARI due to SARS-CoV-2 infection
Test Negative Design Outcome: VE calculated as 1 minus the OR comparing the odds of >2 doses with BNT162b2 for ED cases and controls, multiplied by 100%. | up to three years
  To describe the effectiveness of >2 doses of BNT162b2 against ED admission (without subsequent hospitalization) for ARI due to SARS-CoV-2 infection
Test Negative Design Outcome: BNT162b2 VE estimates stratified by virus variant (as determined by genome sequencing) and select descriptive analyses described above by number of doses received | up to three years
  To further describe the effectiveness of BNT162b2 against hospitalization and ED admission stratified by prevalent or important viral strains
Test Negative Design Outcome: BNT162b2 VE estimates against severe outcomes including ICU admission, mechanical ventilation, and death by number of doses received. | up to three years
  To evaluate the effectiveness of BNT162b2 against severe hospitalization-related outcomes (e.g., ICU admission, mechanical ventilation, and death)
Test Negative Design Outcome: Monthly VE estimates between variants of interest using independent Z tests of log hazard ratios. | up to three years
  To evaluate overall and variant-specific effectiveness of BNT162b2 against SARS-CoV-2 infections and COVID-19 related hospital admissions by time since vaccination (by month)
Test Negative Design Outcome: VE calculated as 1 minus the odds ratio (OR) comparing the odds of being vaccinated with BNT162b2 BA.4/BA.5 bivalent booster for hospitalized cases and controls, multiplied by 100%. | up to three years
  To estimate the effectiveness of the BNT162b2 BA.4/BA.5 bivalent booster against hospitalization for ARI due to SARS-CoV-2 infection.
Test Negative Design Outcome: VE calculated as 1 minus the odds ratio (OR) comparing the odds of being vaccinated with BNT162b2 BA.4/BA.5 bivalent for emergency room admissions/urgent care visit cases and controls, multiplied by 100%. | up to three years
  To estimate the effectiveness of the BNT162b2 BA.4/BA.5 bivalent booster against emergency room admissions/urgent care vists for ARI due to SARS-CoV-2 infection.
Cohort Design Outcome: VE calculated as 1 minus the HR comparing the incidence of 2 doses with BNT162b2 for ED admission due to SARS-CoV-2 infection and not, multiplied by 100%. | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against ED admission (without subsequent hospitalization) ED admission due to SARS-CoV-2 infection
Cohort Design Outcome: VE calculated as 1 minus the HR comparing the incidence of 2 doses with BNT162b2 for ICU admission due to SARS-CoV-2 infection and not, multiplied by 100%. | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against ICU admission due to SARS-CoV-2 infection
Cohort Design Outcome: VE calculated as 1 minus the HR comparing the incidence of (2 doses with BNT162b2 for death due to SARS-CoV-2 infection and not, multiplied by 100%. | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against death due to SARS-CoV-2 infection
Cohort Design Outcome: VE calculated as 1 minus the HR comparing the incidence of 2 doses with BNT162b2 for COVID-19 outpatient visits (without subsequent hospitalization within 14 days) due to SARS-CoV-2 infection and not, multiplied by 100%. | up to three years
  To estimate the effectiveness of 2 doses of BNT162b2 against COVID-19 outpatient visits (without subsequent hospitalization within 14 days) due to SARS-CoV-2 infection
Cohort Design Outcome: VE = 1 minus the HR comparing the incidence of 1 dose of BNT162b2 for hospitalization, ED visit, death, and COVID-19 outpatient visits (without subsequent hosp. within 14 days) due to SARS-CoV-2 and not, multiplied by 100%. | up to three years
  To describe the effectiveness of only 1 dose of BNT162b2 (i.e., partially vaccinated) against hospitalization, ED admission, ICU admission, death, and outpatient visits (without subsequent hospitalization within 14 days) due to SARS-CoV-2 infection
Cohort Design Outcome: VE = 1 minus the HR comparing the incidence ≥1 dose of BNT162b2 (for hospitalization, ED visit, death, and COVID-19 outpatient visits (without subsequent hosp. within 14 days) due to SARS-CoV-2 and not, multiplied by 100%. | up to three years
  To describe the effectiveness of ≥1 dose of BNT162b2 (i.e., ever vaccinated) against hospitalization, ICU admission, ED admission, death, and outpatient visits (without subsequent hospitalization within 14 days) due to SARS-CoV-2 infection
Cohort Design Outcome: VE = 1 minus the HR comparing the incidence of >2 doses of BNT162b2 for hospitalization, ED visit, death, and COVID-19 outpatient visits (without subsequent hosp. within 14 days) due to SARS-CoV-2, multiplied by 100%. | up to three years
  To describe the effectiveness of >2 doses of BNT162b2 against hospitalization, ED admission, ICU admission, death, and outpatient visits (without subsequent hospitalization within 14 days) due to SARS-CoV-2 infection.
XBB.1.5 -adapted monovalent vaccine against critical illness | up to three years
  To describe the effectiveness of XBB.1.5-adapted monovalent vaccine against critical illness (intensive care unit admissions, mechanical ventilation, or inpatient death confirmed by chart review to be COVID-19 related), emergency department, and urgent care visits.
XBB.1.5-adapted monovalent vaccine against outpatient encounters | up to three years
  To describe the effectiveness of XBB.1.5-adapted monovalent vaccine against outpatient encounters.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Tartof SY, Slezak JM, Puzniak L, Hong V, Frankland TB, Ackerson BK, Xie F, Takhar H, Ogun OA, Simmons S, Zamparo JM, Valluri SR, Jodar L, McLaughlin JM. Effectiveness of BNT162b2 BA.4/5 bivalent mRNA vaccine against a range of COVID-19 outcomes in a large health system in the USA: a test-negative case-control study. Lancet Respir Med. 2023 Dec;11(12):1089-1100. doi: 10.1016/S2213-2600(23)00306-5. Epub 2023 Oct 25. PMID 37898148
- [Derived] Tartof SY, Slezak JM, Puzniak L, Hong V, Frankland TB, Xie F, Ackerson BK, Valluri SR, Jodar L, McLaughlin JM. Effectiveness and durability of BNT162b2 vaccine against hospital and emergency department admissions due to SARS-CoV-2 omicron sub-lineages BA.1 and BA.2 in a large health system in the USA: a test-negative, case-control study. Lancet Respir Med. 2023 Feb;11(2):176-187. doi: 10.1016/S2213-2600(22)00354-X. Epub 2022 Oct 7. PMID 36216013
- [Derived] Tartof SY, Slezak JM, Puzniak L, Hong V, Xie F, Ackerson BK, Valluri SR, Jodar L, McLaughlin JM. Durability of BNT162b2 vaccine against hospital and emergency department admissions due to the omicron and delta variants in a large health system in the USA: a test-negative case-control study. Lancet Respir Med. 2022 Jul;10(7):689-699. doi: 10.1016/S2213-2600(22)00101-1. Epub 2022 Apr 22. PMID 35468336
- [Derived] Tartof SY, Slezak JM, Fischer H, Hong V, Ackerson BK, Ranasinghe ON, Frankland TB, Ogun OA, Zamparo JM, Gray S, Valluri SR, Pan K, Angulo FJ, Jodar L, McLaughlin JM. Effectiveness of mRNA BNT162b2 COVID-19 vaccine up to 6 months in a large integrated health system in the USA: a retrospective cohort study. Lancet. 2021 Oct 16;398(10309):1407-1416. doi: 10.1016/S0140-6736(21)02183-8. Epub 2021 Oct 4. PMID 34619098
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591014